CLINICAL TRIAL: NCT00095940
Title: Molecular Biology and Phase II Study of Lapatinib (GW572016) in Pediatric Patients With Recurrent or Refractory Medulloblastoma, Malignant Glioma or Ependymoma
Brief Title: Lapatinib in Treating Young Patients With Recurrent or Refractory Central Nervous System Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-03007; NCI-2012-03007 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PBTC-016 (Other: Pediatric Brain Tumor Consortium); PBTC-016 (Other: CTEP); U01CA081457 (NIH)
Record Dates: First submitted 2004-11-09; First posted 2004-11-09 (Estimated); Results first posted 2012-02-06 (Estimated); Last update posted 2014-05-23 (Estimated); Status verified 2013-01

CONDITIONS: Recurrent Childhood Anaplastic Astrocytoma; Recurrent Childhood Brain Stem Glioma; Recurrent Childhood Ependymoma; Recurrent Childhood Giant Cell Glioblastoma; Recurrent Childhood Glioblastoma; Recurrent Childhood Gliosarcoma; Recurrent Childhood Medulloblastoma; Recurrent Childhood Oligodendroglioma
MeSH Terms: conditions — Astrocytoma; Familial ependymoma; Glioblastoma; Medulloblastoma; Oligodendroglioma | interventions — Lapatinib; N-(3-chloro-4-((3-fluorobenzyl)oxy)phenyl-6-(5-((methylsulfonyl)ethyl)aminomethyl)-2-furyl)-4-quinazolinamine; Magnetic Resonance Spectroscopy; 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole

ARMS (1):
- Treatment (surgery, lapatinib) (Experimental): Molecular Biology Phase: Patients randomized to receive lapatinib prior to surgery receive oral lapatinib twice daily for 7-14 days. Surgery is performed after 7-14 days of lapatinib treatment. For patients randomized to not receive lapatinib, surgery is performed within 3 weeks of registration. After surgical resection, all molecular biology participants start lapatinib treatment within 10 days post-surgery. The first dose of lapatinib post-surgery initiates course 1. Patients receive oral lapatinib twice daily on days 1-28. Treatment repeats every 28 days for up to 26 courses (2 years) in the absence of disease progression or unacceptable toxicity.
  Lapatinib Continuation/Phase II: Patients receive oral lapatinib twice daily on days 1-28. Treatment repeats every 28 days for up to 26 courses (2 years) in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: lapatinib ditosylate; Procedure: therapeutic conventional surgery; Other: laboratory biomarker analysis; Other: pharmacological study; Procedure: positron emission tomography; Procedure: magnetic resonance imaging

INTERVENTIONS:
Drug: lapatinib ditosylate — Given orally
  Other Names: GSK572016; GW-572016; GW2016; Lapatinib; Tykerb
Procedure: therapeutic conventional surgery — Undergo surgery
Other: laboratory biomarker analysis — Correlative studies
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Procedure: positron emission tomography — Correlative studies
  Other Names: FDG-PET; PET; PET scan; tomography, emission computed
Procedure: magnetic resonance imaging — Correlative studies
  Other Names: MRI; NMR imaging; NMRI; nuclear magnetic resonance imaging

SUMMARY:
This phase I/II trial studies lapatinib to see how well it works in treating young patients with recurrent or refractory central nervous system (CNS) tumors. Lapatinib may stop the growth of tumor cells by blocking the enzymes necessary for their growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the MTD and describe the DLT of oral lapatinib (GW572016) administered twice daily for 28 days to children with recurrent or refractory malignant brain tumors who are not receiving steroids (Stratum 1) and to describe toxicities in those who are receiving steroids (Stratum 2).

II. To test the ability of lapatinib (GW572016) to inhibit ERBB receptor signaling in recurrent or refractory: medulloblastoma/PNET, high-grade glioma or ependymomas.

III. To estimate the sustained objective response rates (CR plus PR sustained for 8 weeks) to lapatinib (GW572016) administered continuously at the MTD (900 mg/m2/dose bid) to children with recurrent or refractory: medulloblastoma/PNET, high-grade glioma or ependymoma.

SECONDARY OBJECTIVES:

I. To characterize the plasma pharmacokinetics of lapatinib (GW572016) and tumor tissue lapatinib (GW572016) concentration in children.

II. To assess the effect of steroids on the pharmacokinetics of lapatinib (GW572016).

III. To explore the pharmacogenetic polymorphisms in lapatinib (GW572016) metabolizing enzymes and relate these polymorphisms to the drug pharmacokinetics.

IV. To estimate the incidence of ERBB1, ERBB2, ERBB3 and ERBB4 expression and pathway activation in recurrent or refractory CNS tumors of childhood, including ependymoma, medulloblastoma/PNET and glioma.

V. To identify additional genes both within and outside the canonical ERBB pathway that might act as determinants of response to lapatinib (GW572016).

VI. To explore changes in PET and correlative magnetic resonance imaging in children receiving lapatinib. Imaging studies may be combined across similar PBTC protocols to increase the power for detecting correlations among scans and associations with outcome.

OUTLINE: This is an open-label, multicenter study. Patients are stratified according to histology (medulloblastoma/primitive neuroectodermal tumor vs high-grade glioma vs ependymoma).

Molecular Biology Phase: Patients randomized to receive lapatinib prior to surgery receive oral lapatinib twice daily for 7-14 days. Surgery is performed after 7-14 days of lapatinib treatment. For patients randomized to not receive lapatinib, surgery is performed within 3 weeks of registration. After surgical resection, all molecular biology participants start lapatinib treatment within 10 days post-surgery. The first dose of lapatinib post-surgery initiates course 1. Patients receive oral lapatinib twice daily on days 1-28. Treatment repeats every 28 days for up to 26 courses (2 years) in the absence of disease progression or unacceptable toxicity.

Lapatinib Continuation/Phase II: Patients receive oral lapatinib twice daily on days 1-28. Treatment repeats every 28 days for up to 26 courses (2 years) in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed for at least 30 days.

ELIGIBILITY:
Inclusion Criteria:

* PHASE I TRIAL:

  * All patients with recurrent or refractory malignant CNS tumors; a histological diagnosis of malignant CNS tumor from either the initial presentation or at the time of recurrence is required for all patients, but those with brain stem gliomas

MOLECULAR BIOLOGY TRIAL:

* Patients must have recurrent or refractory disease with a histological diagnosis from either the initial presentation or at the time of recurrence of one of the following:

  * Recurrent or refractory medulloblastoma/PNET
  * Recurrent or refractory high grade glioma, (anaplastic astrocytoma, glioblastoma multiforme, gliosarcoma, anaplastic oligodendroglioma)
  * Recurrent or refractory ependymoma
* Patients for whom surgical resection is clinically indicated and are amenable to receiving GW572016 for 7-14 days prior to their resection

PHASE II TRIAL:

* Patients must have recurrent or refractory disease with a histological diagnosis from either the initial presentation or at the time of recurrence of one of the following:

  * Recurrent or refractory medulloblastoma/PNET,
  * Recurrent or refractory high grade glioma, (anaplastic astrocytoma, glioblastoma multiforme, gliosarcoma, anaplastic oligodendroglioma)
  * Recurrent or refractory ependymoma
* Patients must have measurable disease

  * Patients with neurological deficits should have deficits that are stable for a minimum of 1 week prior to registration
  * Karnofsky performance scale (KPS for > 16 yrs of age) or Lansky performance score (LPS for =< 16 years of age) >= 50 assessed within two weeks prior to registration
  * Evidence of recovery from prior chemotherapy; no myelosuppressive anticancer chemotherapy within 3 weeks and no biological therapy or other non-myelosuppressive investigational agent =< 7 days prior to study registration (6 weeks if a nitrosourea or mitomycin C agent) prior to registration
  * >= 3 months prior to registration for craniospinal irradiation (>= 18 Gy); >= 4 weeks for local radiation to primary tumor; and >= 2 weeks prior to registration for focal irradiation to symptomatic metastatic sites
  * >= 6 months prior to registration for allogeneic bone marrow transplants and >= 3 months prior to registration for autologous bone marrow/stem cell transplants
  * Patients with seizure disorder may be enrolled if well controlled; patients receiving enzyme inducing anticonvulsants are not eligible for this study; patients must be off EIACD for at least 2 weeks prior to registration
  * Patients who are receiving corticosteroids must be on a stable or decreasing dose for at least 1 week prior to registration; patients enrolled in the molecular biology and phase II components of the study will not be stratified based on steroid use; however, use of steroids should be reported as a concomitant medication in the database; in the phase I component of the study, patients on corticosteroids will be eligible for stratum 2 of the study; patients with ACTH deficiency who are on physiological replacement doses of hydrocortisone (or other corticosteroid) will be eligible for stratum 1 of the study
  * Off all colony forming growth factor(s) >= 2 weeks prior to registration (G-CSF, GM-CSF, Erythropoietin)
  * Patients must not have received:
* CYP3A4 inhibitors within seven (7) days prior to registration on protocol and for the duration of the study; however, amiodarone, another CYP3A4 inhibitor, should have been discontinued 6 months prior to registration and for the duration of the study
* CYP3A4 inducers within fourteen (14) days prior to registration and for the duration of the study
* Cimetidine within 48 hours prior to registration and for the duration of the study

  * Patients must be in adequate general condition for study
  * Absolute neutrophil count >= 1000/microliter
  * Platelets >= 100,000/microliter (transfusion independent)
  * Hemoglobin >= 8.0 g/dL (transfusion independent)
  * Serum creatinine =< 1.5 times upper limit of institutional normal for age or GFR >= 70 ml/min/1.73m^2
  * Bilirubin =< 1.5 times upper limit of normal for age
  * SGPT (ALT) < 2.5 x institutional upper limit of normal
  * Albumin >= 2 g/dL
  * No overt renal, hepatic, biliary, cardiac or pulmonary disease
  * Adequate cardiac function, assessed within 2 weeks prior to registration, defined as: shortening fraction of >= 27% by echocardiogram, or ejection fraction >= 50% by gated radionuclide study
  * Adequate pulmonary function, assessed within 2 weeks prior to registration, defined as: no evidence of dyspnea at rest, no exercise intolerance, and a pulse oximetry > 94% if there is clinical indication for determination
  * Patients of childbearing or child fathering potential must be willing to use a medically acceptable form of birth control, which includes abstinence, while being treated on this study
  * Signed informed consent according to institutional guidelines must be obtained

Exclusion Criteria:

* Patients with any significant medical illnesses that, in the investigator's opinion, cannot be adequately controlled with appropriate therapy or would compromise the patient's ability to tolerate this therapy
* Patients with any disease that would obscure toxicity or dangerously alter drug metabolism
* Patients with uncontrolled infection

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 52 (Actual)
Dates: Start 2004-10; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maryam Fouladi, Principal Investigator — Pediatric Brain Tumor Consortium
Locations (1):
- Pediatric Brain Tumor Consortium, Memphis, Tennessee, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants from institutions in the Pediatric Brain Tumor Consortium were enrolled between November 2006 and October 2008.
Pre-assignment Details: Participants with tumors for whom surgical resection was indicated enrolled on the molecular biology phase and randomized to 1) receive lapatinib for 7-14 days pre-surgery or 2) no lapatinib pre-surgery. Those in group 2 who had measurable disease post-surgery would be included in the phase II part as well, but no participant met this criteria.
Groups:
- Medulloblastoma: Lapatinib Prior to Surgery; Ependymoma: Lapatinib Prior to Surgery: Participants with recurrent medulloblastoma who had surgical resection of the tumor at study enrollment and were randomized to receive lapatinib 7-14 days prior to surgery. These participants were not eligible for the phase II objectives.
- Medulloblastoma: No Lapatinib Prior to Surgery: Participants with recurrent medulloblastoma who had surgical resection of the tumor at study enrollment and were randomized to not receive lapatinib prior to surgery. Participants who had measurable disease after surgery were eligible for the phase II objectives.
- Medulloblastoma: No Surgery: Participants with recurrent medulloblastoma who did not have surgical resection of the tumor at study enrollment. These participants contributed to the phase II objectives.
- High Grade Glioma: Lapatinib Prior to Surgery: Participants with recurrent high grade glioma who had surgical resection of the tumor at study enrollment and were randomized to receive lapatinib 7-14 days prior to surgery. These participants were not eligible for the phase II objectives.
- High Grade Glioma: No Lapatinib Prior to Surgery: Participants with recurrent high grade glioma who had surgical resection of the tumor at study enrollment and were randomized to not receive lapatinib 7-14 days prior to surgery. Participants who had measurable disease after surgery were eligible for the phase II objectives.
- High Grade Glioma: No Surgery: Participants with recurrent high grade glioma who did not have surgical resection of the tumor at study enrollment. These participants contributed to the phase II objectives.
- Ependymoma: No Lapatnib Prior to Surgery: Participants with recurrent ependymoma who had surgical resection of the tumor at study enrollment and were randomized to not receive lapatinib 7-14 days prior to surgery. Participants who had measurable disease after surgery were eligible for the phase II objectives.
- Ependymoma: No Surgery: Participants with recurrent ependymoma who did not have surgical resection of the tumor at study enrollment. These participants contributed to the phase II objectives.
Period: Molecular Biology Phase
Arm/Group | Medulloblastoma: Lapatinib Prior to Surgery | Medulloblastoma: No Lapatinib Prior to Surgery | Medulloblastoma: No Surgery | High Grade Glioma: Lapatinib Prior to Surgery | High Grade Glioma: No Lapatinib Prior to Surgery | High Grade Glioma: No Surgery | Ependymoma: Lapatinib Prior to Surgery | Ependymoma: No Lapatnib Prior to Surgery | Ependymoma: No Surgery
Started | 2 | 2 | 0 (No surgery prior to study enrollment; not eligible for the molecular biology phase) | 0 | 0 | 0 (No surgery prior to study enrollment; not eligible for the molecular biology phase) | 2 | 2 | 0 (No surgery prior to study enrollment; not eligible for the molecular biology phase)
Completed | 2 | 2 | 0 | 0 | 0 | 0 | 2 | 2 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Lapatinib Continuation/Phase II
Arm/Group | Medulloblastoma: Lapatinib Prior to Surgery | Medulloblastoma: No Lapatinib Prior to Surgery | Medulloblastoma: No Surgery | High Grade Glioma: Lapatinib Prior to Surgery | High Grade Glioma: No Lapatinib Prior to Surgery | High Grade Glioma: No Surgery | Ependymoma: Lapatinib Prior to Surgery | Ependymoma: No Lapatnib Prior to Surgery | Ependymoma: No Surgery
Started | 2 (Continued to receive lapatinib but were ineligible for the phase II.) | 2 (No measurable disease post surgery - ineligible for the phase II. Continued to receive lapatinib.) | 17 | 0 | 0 | 13 | 2 (Continued to receive lapatinib but were ineligible for the phase II.) | 2 (No measurable disease post surgery - ineligible for the phase II. Continued to receive lapatinib.) | 14
Completed | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Not Completed | 2 | 2 | 16 | 0 | 0 | 13 | 2 | 2 | 13
Not completed — Disease Progression | 1 | 1 | 15 | 0 | 0 | 13 | 2 | 1 | 12
Not completed — Withdrawal by Subject | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Medulloblastoma: Lapatinib Prior to Surgery | Medulloblastoma: No Lapatinib Prior to Surgery | Medulloblastoma: No Surgery | High Grade Glioma: No Surgery | Ependymoma: Lapatinib Prior to Surgery | Ependymoma: No Lapatnib Prior to Surgery | Ependymoma: No Surgery | Total
Number analyzed (Participants) | 2 | 2 | 17 | 13 | 2 | 2 | 14 | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 2 | 12 | 12 | 2 | 2 | 14 | 45
  Between 18 and 65 years | 1 | 0 | 5 | 1 | 0 | 0 | 0 | 7
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.6 (12.0) | 8.7 (.27) | 14.2 (5.9) | 13.5 (4.5) | 7.1 (1.8) | 9.9 (1.8) | 8.0 (4.1) | 11.6 (5.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 9 | 8 | 1 | 0 | 7 | 26
  Male | 1 | 2 | 8 | 5 | 1 | 2 | 7 | 26
Region of Enrollment [Number; unit: participants]
  United States | 2 | 2 | 17 | 13 | 2 | 2 | 14 | 52

OUTCOME MEASURES:

1. Primary Outcome: Relative Phosphorylation of ERBB2 (Molecular Biology Objective)
Description: Lapatinib may be able to control the growth of tumor cells. To assess the ability of lapatinib to block a molecule, the ERBB2 receptor, that signals tumor cells to divide, fresh frozen tissue from the surgical resection is processed by quantitative western blot analysis to assess the phosphorylation of ERBB2. The relative phosphorylation is a ratio of the phosphorylated ERBB2 measured in the tumor normalized to the level of total receptor protein and housekeeping protein. Lower values suggests more inhibition of the ERRB2 receptor signal and a decreased ability for tumor cell division.
Time Frame: 7-14 days after starting therapy and prior to surgery
Population: Participants enrolled on the molecular biology phase (MBP) and who submitted fresh frozen tissue were included in the analysis for this objective. One patient enrolled on the MBP did not provide fresh frozen tissue and was excluded. The sample size required for this objective was not met.
Measure: Median (Full Range); unit: ratio
Groups:
- Lapatinib Prior to Surgery: Participants with recurrent medulloblastoma, high grade glioma, or ependymoma who had surgical resection of the tumor at study enrollment and were randomized to receive lapatinib 7-14 days prior to surgery.
- No Lapatinib Prior to Surgery: Participants with recurrent medulloblastoma, high grade glioma, or ependymoma who had surgical resection of the tumor at study enrollment and were randomized to not receive lapatinib 7-14 days prior to surgery.
Arm/Group | Lapatinib Prior to Surgery | No Lapatinib Prior to Surgery
Number analyzed (Participants) | 4 | 3
ratio | .21 [.03 to .44] | .50 [.05 to 1.66]

2. Primary Outcome: Number of Participants With a Sustained Objective Response (Complete or Partial Response) (Phase II Objective)
Description: A complete response is defined as complete disappearance of all tumor accompanied by a stable or improving neurologic exam, and a partial response is defined as 50% or more reduction in the tumor size by bi-dimensional measurement and a stable or improving neurologic exam. The response must be sustained for at least 8 weeks. The number of patients with a sustained objective response will be reported separately for each of the three disease groups.
Time Frame: From start of therapy until the earliest of disease progression, death or end of the fourth course (recurrent medulloblastoma and recurrent high grade glioma) or end of the sixth course (recurrent ependymoma)
Population: Participants with measureable residual disease who do not receive lapatinib prior to surgery or who do not have surgical resection of the tumor at study enrollment will be assessed for sustained objective response. Participants must have received at least one dose of lapatinib and remain on treatment for the specified time frame to be evaluable.
Measure: Number; unit: Participants
Groups:
- Recurrent Medulloblastoma: Participants with recurrent medulloblastoma who 1)were randomized to not receive lapatinib prior to surgery and had measureable disease after surgical resection or 2) did not have surgical resection of the tumor at study enrollment.
- Recurrent High Grade Glioma: Participants with recurrent high grade glioma who 1)were randomized to not receive lapatinib prior to surgery and had measureable disease after surgical resection or 2) did not have surgical resection of the tumor at study enrollment.
- Recurrent Ependymoma: Participants with recurrent ependymoma who 1)were randomized to not receive lapatinib prior to surgery and had measureable disease after surgical resection or 2) did not have surgical resection of the tumor at study enrollment.
Arm/Group | Recurrent Medulloblastoma | Recurrent High Grade Glioma | Recurrent Ependymoma
Number analyzed (Participants) | 15 | 13 | 13
Participants | 0 | 0 | 0

3. Secondary Outcome: Tumor to Plasma Lapatinib Concentration (Molecular Biology Objective)
Description: For participants randomized to receive lapatinib 7-14 days prior to surgery, plasma samples will be obtained with the first dose of lapatinib prior to surgery. The lapatinib concentration is measured in both the plasma samples and the tumor tissue obtained at surgery. Reported is the concentration of lapatinib observed in the tumor expressed as a percentage of the concentration observed in plasma.
Time Frame: First dose of lapatinib prior to surgery
Population: The analysis population consists of recurrent medulloblastoma, high grade glioma, or ependymoma patients who were randomized to receive lapatinib prior to surgery, consented to the pharmacokinetic studies and received dose 1 of lapatinib.
Measure: Median (Full Range); unit: percent
Arm/Group | Lapatinib Prior to Surgery
Number analyzed (Participants) | 3
percent | 18 [11 to 22]

4. Secondary Outcome: Maximum Concentration of Lapatinib in Plasma (Phase II Objective)
Description: Serial plasma samples for pharmacokinetic studies of lapatinib will be collected from consenting participants with the first dose of course 1.
Time Frame: First dose of lapatinib in course 1
Population: The analysis population consists of participants with recurrent medulloblastoma, high grade glioma, or ependymoma who did not have surgical resection of the tumor at study enrollment, consented to the pharmacokinetic studies, and received the first dose of lapatinib in course 1.
Measure: Median (Full Range); unit: nanogram/milliliter
Groups:
- Lapatinib: No Surgery: Participants with recurrent medulloblastoma, high grade glioma, or ependymoma who 1)were randomized to not receive lapatinib prior to surgery and had measureable disease after surgical resection or 2) did not have surgical resection of the tumor at study enrollment
Arm/Group | Lapatinib: No Surgery
Number analyzed (Participants) | 13
nanogram/milliliter | 5050 [1915 to 10500]

5. Secondary Outcome: Number of Participants With Tumors Expressing Total ERBB2
Description: Total ERBB2 expression is assessed in participants enrolled in both the molecular biology trial and the phase II trial who provided pre-treatment formalin fixed paraffin embedded tumor material. The tumor material is analyzed by immunohistochemistry for expression of total ERBB2. Low, moderate, and intense expression are combined into one group vs. no total ERBB2 expression.
Time Frame: Pre-treatment
Population: Participants from the molecular biology trial or the phase II trial who consented to the biology studies and provided pre-treatment formalin fixed paraffin embedded tumor were included in the analysis population.
Measure: Number; unit: Participants
Groups:
- Recurrent Medulloblastoma: Participants with recurrent medulloblastoma who provided formalin fixed paraffin embedded tumor material prior to treatment were included in the analysis population.
- Recurrent High Grade Glioma: Participants with recurrent high grade glioma who provided formalin fixed paraffin embedded tumor material prior to treatment were included in the analysis population.
- Recurrent Ependymoma: Participants with recurrent ependymoma who provided formalin fixed paraffin embedded tumor material prior to treatment were included in the analysis population.
Arm/Group | Recurrent Medulloblastoma | Recurrent High Grade Glioma | Recurrent Ependymoma
Number analyzed (Participants) | 9 | 7 | 9
Participants | 1 | 2 | 7

6. Secondary Outcome: Number of Participants With Tumors Expressing Phosphorylated ERBB2 (Phase II Objective)
Description: Phosphorylated ERBB2 expression is assessed in patients who provided pre-treatment formalin fixed paraffin embedded tumor material. The tumor material is analyzed by immunohistochemistry for expression of phosphorylated ERBB2. Low, moderate, and intense expression are combined into one group vs. no phosphorylated ERBB2 expression.
Time Frame: Pre-treatment
Population: as for outcome 5
Measure: Number; unit: Participants
Arm/Group | Recurrent Medulloblastoma | Recurrent High Grade Glioma | Recurrent Ependymoma
Number analyzed (Participants) | 9 | 7 | 9
Participants | 1 | 4 | 6

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from day 1 of starting treatment until 30 days after ceasing treatment (off study). AEs possibly, probably, or definitely attributed to the study drug that occured after the off study date were also collected.
Description: One participant in the Medulloblastoma: No Surgery group did not receive any lapatinib as the patient experienced clinical progression prior to starting therapy. This patient is excluded from the adverse event reporting.
Groups:
- Medulloblastoma: Lapatinib Prior to Surgery; Ependymoma: Lapatinib Prior to Surgery: Participants with recurrent medulloblastoma who had surgical resection of the tumor at study enrollment and were randomized to receive lapatinib 7-14 days prior to surgery.
- Medulloblastoma: No Lapatinib Prior to Surgery: Participants with recurrent medulloblastoma who had surgical resection of the tumor at study enrollment and were randomized to not receive lapatinib prior to surgery.
- Medulloblastoma: No Surgery: Participants with recurrent medulloblastoma who did not have surgical resection of the tumor at study enrollment.
- High Grade Glioma: No Surgery: Participants with recurrent high grade glioma who did not have surgical resection of the tumor at study enrollment.
- Ependymoma: No Lapatnib Prior to Surgery: Participants with recurrent ependymoma who had surgical resection of the tumor at study enrollment and were randomized to not receive lapatinib 7-14 days prior to surgery.
- Ependymoma: No Surgery: Participants with recurrent ependymoma who did not have surgical resection of the tumor at study enrollment and were not eligible for the randomization to receive lapatinib or not prior to surgery.
Arm/Group | Medulloblastoma: Lapatinib Prior to Surgery | Medulloblastoma: No Lapatinib Prior to Surgery | Medulloblastoma: No Surgery | High Grade Glioma: No Surgery | Ependymoma: Lapatinib Prior to Surgery | Ependymoma: No Lapatnib Prior to Surgery | Ependymoma: No Surgery
Serious Adverse Events (participants affected / at risk) | 2/2 | 1/2 | 9/16 | 10/13 | 2/2 | 1/2 | 6/14
Other Adverse Events (participants affected / at risk) | 2/2 | 2/2 | 16/16 | 13/13 | 2/2 | 2/2 | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Medulloblastoma: Lapatinib Prior to Surgery (N=2) | Medulloblastoma: No Lapatinib Prior to Surgery (N=2) | Medulloblastoma: No Surgery (N=16) | High Grade Glioma: No Surgery (N=13) | Ependymoma: Lapatinib Prior to Surgery (N=2) | Ependymoma: No Lapatnib Prior to Surgery (N=2) | Ependymoma: No Surgery (N=14)
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
AST,SGOT (serum glutamic oxaloacetic transaminase) (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 2
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ataxia (incoordination) (Nervous system disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 0
Bilirubin (hyperbilirubinemia) (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fever (in the absence of neutropenia) (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Leak, cerebrospinal fluid (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Leukocytes (Investigations) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Lymphopenia (Investigations) | 0 | 0 | 3 | 3 | 0 | 0 | 1
Neutrophils/granulocytes (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 1 | 0 | 3 | 1 | 0 | 0 | 1
Platelets (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 1 | 1 | 2
Seizure (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 2
Somnolence/depressed level of consciousness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Speech impairment (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Medulloblastoma: Lapatinib Prior to Surgery (N=2) | Medulloblastoma: No Lapatinib Prior to Surgery (N=2) | Medulloblastoma: No Surgery (N=16) | High Grade Glioma: No Surgery (N=13) | Ependymoma: Lapatinib Prior to Surgery (N=2) | Ependymoma: No Lapatnib Prior to Surgery (N=2) | Ependymoma: No Surgery (N=14)
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 0 | 1 | 4 | 4 | 0 | 1 | 7
AST, SGOT (serum glutamic oxaloacetic transaminase) (Investigations) | 0 | 2 | 1 | 4 | 0 | 0 | 5
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 1 | 0 | 1 | 3 | 0 | 1 | 4
Alkaline phosphatase (Investigations) | 0 | 1 | 0 | 1 | 0 | 1 | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1
Amylase (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 2 | 4 | 2 | 1 | 1 | 1
Ataxia (Nervous system disorders) | 0 | 0 | 2 | 2 | 0 | 0 | 2
Bicarbonate, serum-low (Metabolism and nutrition disorders) | 0 | 0 | 2 | 1 | 1 | 1 | 4
Bilirubin (hyperbilirubinemia) (Investigations) | 0 | 1 | 4 | 2 | 2 | 0 | 4
Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 0 | 0 | 4 | 3 | 1 | 1 | 2
Cholesterol, serum-high (hypercholesteremia) (Investigations) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Confusion (Psychiatric disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 3
Creatinine (Investigations) | 0 | 0 | 1 | 2 | 0 | 0 | 0
Cushingoid appearance (Endocrine disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Cystitis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 3 | 0 | 1 | 0 | 2
Diarrhea (Gastrointestinal disorders) | 2 | 2 | 13 | 7 | 2 | 1 | 12
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 2 | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 3 | 1 | 0 | 1 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Enteritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Extremity-upper (function) (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fever (in the absence of neutropenia) (General disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 5
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
GGT (gamma-Glutamyl transpeptidase) (Investigations) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 0 | 0 | 2 | 3 | 1 | 1 | 5
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 0 | 0 | 4 | 0 | 1 | 1 | 2
Hair loss/alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1
Heartburn/dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hydrocephalus (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Incontinence, anal (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Incontinence, urinary (Renal and urinary disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Irritability (children < 3 years of age) (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Leak, cerebrospinal fluid (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Leukocytes (Investigations) | 0 | 2 | 5 | 1 | 2 | 0 | 1
Lymphopenia (Investigations) | 1 | 0 | 7 | 5 | 1 | 1 | 2
Magnesium, serum-high (hypermagnesemia) (Metabolism and nutrition disorders) | 0 | 0 | 1 | 3 | 1 | 0 | 0
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 0 | 0 | 3 | 0 | 0 | 0 | 1
Nail changes (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 3 | 0 | 1 | 0 | 5
Neutrophils/granulocytes (Investigations) | 0 | 1 | 0 | 1 | 0 | 0 | 1
Nystagmus (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ophthalmoplegia/diplopia (double vision) (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Personality/behavioral (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 0 | 1 | 4 | 3 | 1 | 1 | 6
Platelets (Investigations) | 0 | 0 | 2 | 0 | 1 | 0 | 0
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 2
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 0 | 0 | 4 | 5 | 2 | 0 | 4
Proteinuria (Renal and urinary disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 1
Pruritus/itching (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rash/desquamation (Skin and subcutaneous tissue disorders) | 0 | 2 | 3 | 1 | 0 | 0 | 7
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 3 | 2 | 0 | 0 | 1
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 0
Sodium, serum-high (hypernatremia) (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 0 | 0 | 1 | 2 | 1 | 0 | 2
Somnolence/depressed level of consciousness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Speech impairment (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Sweating (diaphoresis) (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Triglyceride, serum-high (hypertriglyceridemia) (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1
Urinary frequency/urgency (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Urine color change (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Vision-photophobia (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Voice changes/dysarthria (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 9 | 4 | 0 | 1 | 7
Weight loss (Investigations) | 0 | 2 | 2 | 1 | 0 | 0 | 0
Extremity-lower (gait/walking) (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2

LIMITATIONS AND CAVEATS:
Accrual to the Molecular Biology phase (MBP) was contingent upon accrual being open for the Phase II since some participants in the MBP could be counted in the phase II. The phase II enrolled rapidly thus limiting enrollment to the MBP.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less